CLINICAL TRIAL: NCT06766539
Title: The Application of Eye-Tracking Technology in Perioperative Management and Education: a Prospective Observational Study
Brief Title: The Application of Eye-Tracking Technology in Perioperative Management and Education
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1282
Record Dates: First submitted 2024-12-22; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Eye-tracking Technology; Medical Education; Perioperative Management; Attention Distribution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore the value of eye-tracking technology in perioperative management and teaching. The study aims to understand how eye-tracking can help analyze the attention distribution of clinicians during perioperative procedures and optimize workflows for improved safety and teaching outcomes.

The main questions it seeks to answer are:

How does eye-tracking technology reveal the focus distribution patterns of experienced and novice clinicians in perioperative scenarios? Can visualizing expert clinicians' eye movement patterns improve the learning outcomes and operational skills of medical students?

Participants include anesthesiologists and medical students involved in perioperative management training. Eye-tracking data, such as fixation duration, fixation count, and heatmaps, will be collected during surgical and training scenarios. The study will analyze correlations between attention distribution and operational performance. This research will provide insights into optimizing perioperative safety and revolutionizing medical education using objective attention data.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists, including senior physicians and junior doctors.
* Medical students undergoing perioperative management training.

Exclusion Criteria:

* Individuals with ophthalmological conditions that affect eye movement function.
* Participants who fail to complete the full experimental protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiologists, including senior physicians and junior doctors and medical students undergoing perioperative management training.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identify the "hotspots" where anesthesiologists focus their attention within different areas of the anesthesia machines. | 1 year
  Every anesthesiologist will record data from three cases. Data collection will commence as the general anesthesia procedure begins when the patient moves onto the surgical table and will complete when the patient reaches the states of sedation and unconsciousness in preparation for the operation. This period, during which the anesthesiologist plays a leading role, typically lasts less than 10 minutes. No data will be recorded once the surgical operation begins.
  The Tobii eye-tracker will generate a diverse dataset, encompassing eye trajectory, fixation (a gaze resting on a spot for more than 150 ms), saccades (rapid eye movements between two distinct points), and pupil size. This comprehensive dataset enables us to identify the "hotspots" where anesthesiologists focus their attention within different areas of the anesthesia machines.

SECONDARY OUTCOMES:
The percentage of time anesthesiologists' eyes attention. | 1 year
  Moreover, we will calculate the percentage of time anesthesiologists' eyes spend on team members. We will also quantify the duration of eye contact and communication content between the anesthesiologist and each team member.
Attention of the clinician | 1 year
  Finally, we will examine the correlation between these behavioral measures (e.g., fixation on hotspots, percentage of time focused on team members, communication episodes) and the duration of the anesthesia procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China